CLINICAL TRIAL: NCT04275596
Title: Impact of Topical Antiadhesion Therapy on Wound Healing and Postoperative Pain After Anal Surgery: A Randomized Double-blinded Controlled Study
Brief Title: Impact of Topical Antiadhesion Therapy on Wound Healing and Postoperative Pain After Anal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mansoura 123
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Anal Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2QR complex (Active Comparator): Patients who undergo anal surgery will apply 2QR complex topical agent on the wound until healing
  Interventions: Drug: 2QR complex
- Placebo (Active Comparator): Patients who undergo anal surgery will apply placebo cream on the wound until healing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2QR complex — Application of topical gel containing 2QR complex on the anal wound until complete wound healing
  Arms: 2QR complex
Drug: Placebo — Application of topical placebo on the anal wound until complete wound healing
  Arms: Placebo

SUMMARY:
2QR-complex is a patented molecule extracted from Aloe vera barbadensis leaves that blocks the adhesion of pathogenic microbes to human epithelial cells and tissues [9]. Anti-adhesion therapy such as 2QR-complex has been suggested as an alternative to antibiotics in the treatment of bacterial infections. 2QR-complex based products have already shown comparable efficacy to antibiotics in treating mucosal infections such as bacterial vaginosis.

In the present study we aim to assess the efficacy of 2QR-complex in pain relief and promotion of anal wound healing after anal surgery. We presumed that anal discomfort and prolonged healing after surgery for anal fissure, fistula, and hemorrhoids may in part be due to contamination of the wound with fecal bacteria that colonize at the surgical site. Therefore, we assumed that the use of topical anti-adhesive 2QR-complex-based product may serve to minimize this negative impact on wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex with simple anal fistula, chronic anal fissure, or grade III/IV hemorrhoids will be included.

Exclusion Criteria:

* Patients with other anal conditions, diabetic patients, patients under steroid or immunosuppressive therapy will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to complete anal Wound healing | Six weeks after surgery
  The time required to achieve complete Complete epithelization of the anal wound postoperatively

SECONDARY OUTCOMES:
Anal pain | one week, one month, two months after surgery
  pain assessed using visual analogue scale from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided